CLINICAL TRIAL: NCT04535791
Title: Efficacy of Vitamin D Supplementation to Prevent the Risk of Acquiring or Evolving Into the Severe Form of COVID-19 in Healthcare Workers Caring for Patients With the Disease. Blinded Randomized Clinical Trial
Brief Title: Efficacy of Vitamin D Supplementation to Prevent the Risk of Acquiring COVID-19 in Healthcare Workers
Acronym: COVID-19
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Coordinación de Investigación en Salud, Mexico (Other Government)
Collaborators: Hospital Infantil de Mexico Federico Gomez (Other)
Responsible Party: Principal Investigator, Miguel Angel Villasis Keever, Clinical Professor, Coordinación de Investigación en Salud, Mexico
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: R-2020-785-090
Record Dates: First submitted 2020-07-30; First posted 2020-09-02 (Actual); Last update posted 2021-12-22 (Actual); Status verified 2021-12

CONDITIONS: Covid19; Vitamin D
MeSH Terms: conditions — COVID-19 | interventions — Cholecalciferol; Vitamin D

STUDY DESIGN:
Intervention Model Description: Blinded randomized clinical trial
Who Masked: Participant, Care Provider, Investigator
Masking Description: To ensure that participants are unaware of the intervention they are receiving, both the capsules containing vitamin D3 and the placebo will be the same. Cholecalciferol (Vitamin D3), 4000UI tablets will be purchased from the MEDIX laboratory (trade name HISTOFIL). The placebo will consist of corn starch, which will be purchased from a supplier, who packages it in a 25 kg bag. As it is a dry product, the supplier guarantees that the corn starch maintains its characteristics for 3 years, as long as it is stored in closed container, in a cool and dry place, free of moisture, dust, insects and rodents. The encapsulation of the placebo and vitamin D3 will be carried out by an external supplier with capsules of the capsugel brand, maintaining quality control to avoid contamination of the product during storage and encapsulation. An external researcher will have a list to which group each subject belongs, without being in contact with the research.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- cholecalciferol (Vitamin D) (Experimental): cholecalciferol 4,000 IU orally daily (1 capsule) for 30 days
  Interventions: Drug: Cholecalciferol
- Starch (Placebo Comparator): Starch 500 mg orally daily (1 capsule) for 30 days
  Interventions: Drug: Cholecalciferol

INTERVENTIONS:
Drug: Cholecalciferol — 4,000 IU orally daily for 30 days
  Other Names: vitamin D

SUMMARY:
In a blinded randomized clinical trial, which will include health workers (doctors, residents, nurses, stretcher-bearers, technicians, hygiene and cleaning) who are members of the health teams that care for patients with COVID-19. Two groups will be formed: the Vitamin D group taking 4,000 IU orally daily for 30 days, the control group being given a placebo during the same time period.

Participants will be adults, who have not had COVID-19 disease, and who sign the informed consent. At the beginning of the study anthropometric variables (weight, height, BMI) will be taken, the short medical history can be identified to identify comorbidities, and a fasting blood sample will be taken to determine changes in Vitamin D (25 (OH) Vitamin D), in addition to RT-PCR saliva samples, as well as detection of serum antibodies to determine whether or not they have SARS-CoV-2 disease. Participants will follow each other 45 days. Those with COVID-19 disease will be monitored frequently to determine the course of the disease. At the end of 45 days, new samples will be taken to determine levels of vitamin D and antibodies against SARS-Cov-2.

DETAILED DESCRIPTION:
In a blinded randomized clinical trial, which will include health workers (doctors, residents, nurses, stretcher-bearers, technicians, hygiene and cleaning) who are members of the health teams that care for patients with COVID-19. Participants with a history of having COVID-19 disease or who are consuming vitamin D at that time will be excluded. Through randomization, two groups will be formed: the Vitamin D group taking 4,000 IU orally daily for 30 days, the control group being given a placebo (starch) during the same time period. Participants and researchers will be blinded regarding the maneuver.

At the beginning of the study anthropometric variables (weight, height, BMI) will be taken, the short medical history can be identified to identify comorbidities such as diabetes mellitus, hypertension or obesity, and a fasting blood sample will be taken to determine the changes in Vitamin D (25 (OH) VD), in addition to saliva samples by RT-PCR, as well as detection of antibodies in serum to determine whether or not they have SARS-CoV-2 disease. Participants who test positive for COVID-19 will be eliminated by the RT-PCR test. Participants will follow each other 45 days. Contacted weekly to verify the consumption of the capsules, as well as evaluation of adverse effects of vitamin D. Monitored for suspicious data of COVID-19 and in case of presenting the disease by COVID-19, a study will be carried out to confirm the infection through RT-PCR and will be monitored to determine the course of the disease. At the end of 45 days, new samples will be taken to determine levels of vitamin D and antibodies against SARS-Cov-2.

ELIGIBILITY:
Inclusion Criteria:

* Health workers in areas of care for patients with COVI-19
* Adults
* Men and women.
* That they agree to participate in the study by signing the letter of informed consent

Exclusion Criteria:

* Those who know that they have already suffered from COVID-19
* Those who have received a vitamin D supplement in the previous two weeks.
* Difficulty obtaining blood samples

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 321 (Actual)
Dates: Start 2020-07-15 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2021-07-15 (Actual)

PRIMARY OUTCOMES:
Number of Participants with COVID-19 | 45 days
  cases confirmed by RT-PCR for SARS-CoV-2, or by antibody detection.
Number of Participants with hospitalization for COVID-19 | 45 days
  participants who, having developed SARS-CoV-2 infection, require hospitalization for the same condition.

SECONDARY OUTCOMES:
Serum concentration of 25 (OH) vitamin D | the beginning and through study completion, an average of 45 days
  Serum concentration of 25 (OH) vitamin D at the beginning and through study completion, an average of 45 days

CONTACTS AND LOCATIONS:
Overall Officials: Miguel Angel Villasis-Keever, Principal Investigator — Coordinación de Investigación en Salud, Mexico
Locations (1):
- Hospital Centro Medico Nacional Siglo XXI, Mexico City, Mexico City, Mexico

REFERENCES:
- [Derived] Villasis-Keever MA, Lopez-Alarcon MG, Miranda-Novales G, Zurita-Cruz JN, Barrada-Vazquez AS, Gonzalez-Ibarra J, Martinez-Reyes M, Grajales-Muniz C, Santacruz-Tinoco CE, Martinez-Miguel B, Maldonado-Hernandez J, Cifuentes-Gonzalez Y, Klunder-Klunder M, Garduno-Espinosa J, Lopez-Martinez B, Parra-Ortega I. Efficacy and Safety of Vitamin D Supplementation to Prevent COVID-19 in Frontline Healthcare Workers. A Randomized Clinical Trial. Arch Med Res. 2022 Jun;53(4):423-430. doi: 10.1016/j.arcmed.2022.04.003. Epub 2022 Apr 18. PMID 35487792